CLINICAL TRIAL: NCT01359956
Title: Fotemustine and Dacarbazine Versus Dacarbazine +/- Alpha Interferon in Advanced Malignant Melanoma: Phase III Study
Brief Title: Fotemustine and Dacarbazine Versus Dacarbazine +/- Alpha Interferon in Advanced Malignant Melanoma
Acronym: SICOG 0109
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SICOG 0109
Record Dates: First submitted 2011-05-13; First posted 2011-05-25 (Estimated); Results first posted 2020-11-13 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2020-09

CONDITIONS: Malignant Melanoma; Recurrent Melanoma
MeSH Terms: conditions — Melanoma | interventions — Dacarbazine; fotemustine; Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A1 (Experimental): combination chemotherapy without interferon
  Interventions: Drug: Dacarbazine; Drug: Fotemustine
- A2 (Experimental): combination chemotherapy with interferon
  Interventions: Drug: Dacarbazine; Drug: Fotemustine; Drug: Interferon Alfa-2b
- B1 (Active Comparator): single agent dacarbazine without interferon
  Interventions: Drug: Dacarbazine
- B2 (Experimental): single agent dacarbazine plus interferon
  Interventions: Drug: Dacarbazine; Drug: Interferon Alfa-2b

INTERVENTIONS:
Drug: Dacarbazine — 900 mg / m2 every 3 weeks
Drug: Fotemustine — 100 mg / m2 every 3 weeks
  Arms: A1; A2
Drug: Interferon Alfa-2b — 5 M units every 3 weeks
  Arms: A2; B2

SUMMARY:
This study evaluated two chemotherapy regimens with and without the addition of interferon in patients with advanced or recurrent melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of malignant melanoma in advanced stage or recurrent after surgery, and not amenable to further surgery or local therapy.
* Presence of measurable disease
* Age > or = 18 years and < or = 75 years
* Performance status (ECOG) 0 - 2 (Appendix 2)
* Life expectancy ³ 3 months
* Adequate bone marrow function (ANC ³ 2,000/mmc; PTL ³ 100,000/mmc; Hb ³ 10 gr/dl), normal liver and renal function (bilirubin < 1.25 x N, creatinine < 1.25 x N, SGOT, SGPT < 3 times upper normal limit of testing laboratory.
* Written, informed consent prior to study specific procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.
* Prior surgery > 3 weeks from initiating .
* If palliative radiation is needed, in case of non target lesions, it must be given prior to initiating chemotherapy. If palliative radiation is required during the study the patient should be permanently discontinued from further treatment.
* Adequate contraceptive measures during study participation for sexually active patients of child bearing potential must implement.

Exclusion Criteria:

* Previous or concurrent malignancies at other sites with the exception of surgically cured carcinoma in-site of the cervix and basal or squamous cell carcinoma of the skin.
* Prior chemo-immunotherapy ( previous adjuvant immunotherapy is allowed)
* Known HIV disease.
* Concurrent treatment with other experimental drugs.
* Concurrent chemotherapy, immunotherapy, hormonal therapy (excluding contraceptives and replacement steroids), radiation therapy
* Pregnant or lactating females Previous or concurrent malignancies at other sites with the exception of surgically cured carcinoma in-site of the cervix and basal or squamous cell carcinoma of the skin.

Prior chemo-immunotherapy ( previous adjuvant immunotherapy is allowed) Known HIV disease. Concurrent treatment with other experimental drugs. Concurrent chemotherapy, immunotherapy, hormonal therapy (excluding contraceptives and replacement steroids), radiation therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2002-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo A Ascierto, M.D., Ph.D., Principal Investigator — NCI Naples; Antonio Daponte, M.D., Principal Investigator — NCI Naples; Simona Signoriello, M.D., Principal Investigator — University of Campania Luigi Vanvitelli

REFERENCES:
- [Result] Daponte A, Signoriello S, Maiorino L, Massidda B, Simeone E, Grimaldi AM, Caraco C, Palmieri G, Cossu A, Botti G, Petrillo A, Lastoria S, Cavalcanti E, Aprea P, Mozzillo N, Gallo C, Comella G, Ascierto PA; Southern Italy Cooperative Oncology Group (SICOG). Phase III randomized study of fotemustine and dacarbazine versus dacarbazine with or without interferon-alpha in advanced malignant melanoma. J Transl Med. 2013 Feb 13;11:38. doi: 10.1186/1479-5876-11-38. PMID 23402397

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomly assigned to one of four treatment groups. Patients were randomized through a computerized procedure of permuted blocks centralized at the coordinating center (Medical Oncology, NCI Napoli), stratified by PS (0-1,2) and site of metastases (visceral, not visceral).
Groups:
- A1 - Combination Chemotherapy Without Interferon: combination chemotherapy without interferon
  Fotemustine: 100 mg / m2 IV on day 1 repeated on a 3 week cycle
  Dacarbazine: 900 mg / m2 IV on day 2 repeated on a 3 week cycle
- A2 - Combination Chemotherapy With Interferon: combination chemotherapy with interferon
  Fotemustine: 100 mg / m2 IV on day 1 repeated on a 3 week cycle
  Dacarbazine: 900 mg / m2 IV on day 2 repeated on a 3 week cycle
  Interferon Alfa-2b: α2b 5 MUI three times per week
- B1 - Single Agent Dacarbazine Without Interferon: single agent dacarbazine without interferon
  Dacarbazine: 900 mg/m2 IV on day 1 repeated on a three-week cycle
- B2 - Single Agent Dacarbazine Plus Interferon: single agent dacarbazine plus interferon
  Dacarbazine: 900 mg / m2 every 3 weeks
  Interferon Alfa-2b: α2b 5 MUI three times per week
Period: Overall Study
Arm/Group | A1 - Combination Chemotherapy Without Interferon | A2 - Combination Chemotherapy With Interferon | B1 - Single Agent Dacarbazine Without Interferon | B2 - Single Agent Dacarbazine Plus Interferon
Started | 67 | 69 | 71 | 62
Completed | 6 | 5 | 4 | 4
Not Completed | 61 | 64 | 67 | 58
Not completed — Death | 58 | 60 | 66 | 57
Not completed — Lost to Follow-up | 3 | 4 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A1 - Combination Chemotherapy Without Interferon | A2 - Combination Chemotherapy With Interferon | B1 - Single Agent Dacarbazine Without Interferon | B2 - Single Agent Dacarbazine Plus Interferon | Total
Number analyzed (Participants) | 64 | 68 | 70 | 58 | 260
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (13) | 50 (15) | 59 (15) | 56 (14) | 55 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 33 | 28 | 20 | 103
  Male | 42 | 35 | 42 | 38 | 157
Region of Enrollment [Number; unit: participants]
  Italy | 64 | 68 | 70 | 58 | 260
Nodular melanoma [Count of Participants; unit: Participants] | 27 | 36 | 36 | 31 | 130

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall Survival was defined as the time from the date of randomisation to the date of death from any cause or the date of last follow-up for living patients.
  OS curves were estimated with the Kaplan - Meier (K-M) method and treatments were compared with a two - sided log - rank test.
Time Frame: 24 months
Population: Nine patients were lost to follow-up immediately after randomization and, in particular, for FDI + FD 132, instead of 136 randomized (4 lost pts.), for DI + D, 128 instead of 133 (5 lost pts.), for FD1 + DI 126, instead of 131 (5 lost pts.), 134 instead of 138 (4 lost pts.)
Measure: Median (Full Range); unit: Months
Groups:
- Fotemustine/Dacarbazine/Interferon + Fotemustine/Dacarbazine: combination chemotherapy with interferon
  Fotemustine: 100 mg / m2 IV on day 1 repeated on a 3 week cycle
  Dacarbazine: 900 mg / m2 IV on day 2 repeated on a 3 week cycle
  Interferon Alfa-2b: α2b 5 MUI three times per week
  combination chemotherapy without interferon
  Fotemustine: 100 mg / m2 IV on day 1 repeated on a 3 week cycle
  Dacarbazine: 900 mg / m2 IV on day 2 repeated on a 3 week cycle
- Dacarbazine/Interferon + Dacarbazine: single agent dacarbazine plus interferon
  Dacarbazine: 900 mg / m2 every 3 weeks
  Interferon Alfa-2b: α2b 5 MUI three times per week
  single agent dacarbazine without interferon
  Dacarbazine: 900 mg/m2 IV on day 1 repeated on a three-week cycle
- Fotemustine/Dacarbazine/Interferon+Dacarbazine/Interferon: combination chemotherapy with interferon
  Fotemustine: 100 mg / m2 IV on day 1 repeated on a 3 week cycle
  Dacarbazine: 900 mg / m2 IV on day 2 repeated on a 3 week cycle
  Interferon Alfa-2b: α2b 5 MUI three times per week
  single agent dacarbazine plus interferon
  Dacarbazine: 900 mg / m2 every 3 weeks
  Interferon Alfa-2b: α2b 5 MUI three times per week
- Fotemustine/Dacarbazine + Dacarbazine: combination chemotherapy without interferon
  Fotemustine: 100 mg / m2 IV on day 1 repeated on a 3 week cycle
  Dacarbazine: 900 mg / m2 IV on day 2 repeated on a 3 week cycle
  single agent dacarbazine without interferon
  Dacarbazine: 900 mg/m2 IV on day 1 repeated on a three-week cycle
Arm/Group | Fotemustine/Dacarbazine/Interferon + Fotemustine/Dacarbazine | Dacarbazine/Interferon + Dacarbazine | Fotemustine/Dacarbazine/Interferon+Dacarbazine/Interferon | Fotemustine/Dacarbazine + Dacarbazine
Number analyzed (Participants) | 132 | 128 | 126 | 134
Months | 7.9 [6.6 to 10.2] | 8.6 [6.3 to 10.4] | 9.1 [6.3 to 11.1] | 7.7 [6.3 to 9.7]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival (PFS) was defined as the time from the date of randomisation to the date of progression of disease or death from any cause, whichever occurred first, or date of last follow-up for patients without progression and alive at the end of the study.
  PFS curves were estimated with the Kaplan - Meier (K-M) method and treatments were compared with a two-sided log-rank test.
Time Frame: 12 months
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | Fotemustine/Dacarbazine/Interferon + Fotemustine/Dacarbazine | Dacarbazine/Interferon + Dacarbazine | Fotemustine/Dacarbazine/Interferon+Dacarbazine/Interferon | Fotemustine/Dacarbazine + Dacarbazine
Number analyzed (Participants) | 132 | 128 | 126 | 134
Months | 2.7 [2.4 to 3.8] | 2.5 [2.3 to 3.7] | 2.8 [2.4 to 3.9] | 2.5 [2.3 to 2.9]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall Response Rate (ORR) included Complete Response (CR) and Partial Response (PR).
  Complete Response (CR) was defined as disappearance of all symptoms and signs of all measurable disease, lasting for at least four weeks, without appearance of new lesions.
  Partial Response (PR) was defined as a > 50% reduction in the sum of the products of the perpendicular diameters of all measurable lesions, lasting for at least four weeks, without appearance of new lesions or enlargement of existing lesions.
Time Frame: 18 weeks from start of therapy
Population: Nine patients were lost to follow-up immediately after randomization and, in particular, for FDI + FD 132, instead of 136 randomized (4 lost pts.), for DI + D 128, instead of 133 (5 lost pts.), for FD1 + DI 126, instead of 131 (5 lost pts.), 134, instead of 138 (4 lost pts.).
Measure: Number; unit: participants
Arm/Group | Fotemustine/Dacarbazine/Interferon + Fotemustine/Dacarbazine | Dacarbazine/Interferon + Dacarbazine | Fotemustine/Dacarbazine/Interferon+Dacarbazine/Interferon | Fotemustine/Dacarbazine + Dacarbazine
Number analyzed (Participants) | 132 | 128 | 126 | 134
participants | 32 | 33 | 34 | 31

4. Secondary Outcome: Treatment Related Toxicity
Description: worst grade CTC toxicity, for each cycle and overall, will be reported for each treatment arm
Time Frame: at end of each 3 week cycle of therapy up to the discontinuation
Population: It wasn't possible to assess the treatment related toxicity for all the patients included in the study because for some of them, no data were collected.
  It's difficult to indicate the exact number of participants affected by the worst grade CTC toxicity because the same patient could be affected by one or more side effects.
Measure: Count of Participants; unit: Participants
Arm/Group | Fotemustine/Dacarbazine/Interferon + Fotemustine/Dacarbazine | Dacarbazine/Interferon + Dacarbazine | Fotemustine/Dacarbazine/Interferon+Dacarbazine/Interferon | Fotemustine/Dacarbazine + Dacarbazine
Number analyzed (Participants) | 129 | 122 | 119 | 132
Participants | 129 | 122 | 119 | 132

ADVERSE EVENTS:
Arm/Group | A1 - Combination Chemotherapy Without Interferon | A2 - Combination Chemotherapy With Interferon | B1 - Single Agent Dacarbazine Without Interferon | B2 - Single Agent Dacarbazine Plus Interferon
Serious Adverse Events (participants affected / at risk) | 14/62 | 27/67 | 8/71 | 10/52
Other Adverse Events (participants affected / at risk) | 12/62 | 25/67 | 16/71 | 13/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A1 - Combination Chemotherapy Without Interferon (N=62) | A2 - Combination Chemotherapy With Interferon (N=67) | B1 - Single Agent Dacarbazine Without Interferon (N=71) | B2 - Single Agent Dacarbazine Plus Interferon (N=52)
Neutropenia (Blood and lymphatic system disorders) | 9 (62) | 27 (67) | 8 (72) | 10 (52)
Platelets (Blood and lymphatic system disorders) | 14 (62) | 23 (67) | 3 (72) | 4 (52)
Anaemia (Blood and lymphatic system disorders) | 4 (62) | 13 (67) | 1 (72) | 2 (52)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A1 - Combination Chemotherapy Without Interferon (N=62) | A2 - Combination Chemotherapy With Interferon (N=67) | B1 - Single Agent Dacarbazine Without Interferon (N=71) | B2 - Single Agent Dacarbazine Plus Interferon (N=52)
Nausea/Vomiting (Gastrointestinal disorders) | 12 | 25 | 16 | 13
Diarrhoea (Gastrointestinal disorders) | 3 | 5 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No